CLINICAL TRIAL: NCT02139085
Title: A Prospective Double Blind Randomized Controlled Trial Of Electrocoagulation Versus Radiofrequency Treatment Of The Great Saphenous Vein In Patients With Varicose Veins.
Brief Title: Great Saphenous Vein Electrocoagulation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Fabio H Rossi, vascular surgeon PhD, Instituto Dante Pazzanese de Cardiologia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IDPC 2014
Record Dates: First submitted 2014-05-12; First posted 2014-05-15 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Venous Disease; Varicose Veins
Keywords: varicose veins; catheter ablation; Catheter Ablation, Electrical; Catheter Ablation, Radiofrequency
MeSH Terms: conditions — Varicose Veins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- GSV Electrocoagulation (Active Comparator): GSV Electrocoagulation Source: Electrosurgical Generator(FX-Valley Lab; USA) Energy: 60 Watts x 10 seconds
  Interventions: Device: GSV Electrocoagulation
- GSV Radiofrequency (Active Comparator): GSV Radiofrequency Source: Closure FAST(Covidien, USA) Energy: 60 Joules / cm
  Interventions: Device: GSV Radiofrequency

INTERVENTIONS:
Device: GSV Electrocoagulation — The energy source will be the Electrosurgical Generator (FX-Valley Lab; USA) and the GSV thermo ablation will be performed with 60 Watts per 10 seconds. The catheter and electrocoagulation device head will be pulled back in increments of 2 cm also to overlap the treatment sites.
  Arms: GSV Electrocoagulation
Device: GSV Radiofrequency — The second generation RF device (Closure FAST; Covidien, USA) will be used. The treatment component of the device is 7 cm in length and works with a segmental pullback protocol. Once the catheter is in position, activation of the generator delivers 20- seconds cycles of energy to the catheter tip, which heats the vein wall to 120 o C.
  Arms: GSV Radiofrequency

SUMMARY:
Introduction: Lower extremity Chronic Venous Insufficiency is a prevalent disease that adversely affects an individual's Quality of Life. Varicose vein endovenous radiofrequency treatment have a lower risk of iatrogenic injuries and offer faster return to work activities, when compared with open surgical techniques. Endovenous electrocoagulation can selectively and safely cause Great Saphenous Vein (GSV) wall necrosis but its clinical results has never been studied before.

Objective: The objective of this study is to compare Great Saphenous Vein electrocoagulation and radio frequency (RF) endovascular varicose vein treatment clinical results and quality of life improvement in a prospective double blind randomized controlled clinical trial.

Methods: Consecutive patients with varicose veins and primary GSV reflux will be randomized to Electrocoagulation or Radiofrequency endovenous treatment. The primary outcome measure will be GSV occlusion rate at 3 and 6 months after treatment verified by Duplex Scanning (DS). Secondary outcome measures will be pain visual analogue scale (VAS), bruising, neuropathy and vein thrombosis frequency in the immediate postoperative period (1 week); and Clinical Etiology Anatomy and Pathophysiology (CEAP) classification ,Venous Clinical Severity Scale (VCSS), and Aberdeen Varicose Vein Questionnaire (AVVQ), obtained preoperatively, at 3 and 6 months postoperatively. For statistical analysis, we will use the Student's t test, the Mann-Whitney test and Pearson's correlation, considering positive statistical significance when level of p <0.05.

DETAILED DESCRIPTION:
All patients included in the study will be preoperatively examined to evaluate the severity of venous disease, using the CEAP classification, VCSS and AVVQ. They will undergo venous DS with the aim of investigating GSV insufficiency, its caliber and depth and presence of previous thrombophlebitis.

Patients will be randomized on the day of surgery with an electronic table of random numbers:

Group 1:Electrocoagulation treatment. Group 2: Radiofrequency treatment.

Patients and outcomes assessor will be blinded to the group of endovenous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic varicose veins of the lower limbs and partial or total failure (venous reflux) of the GSV

Exclusion Criteria:

* Previous varicose vein surgery with removal of the GSV
* Pregnant women
* Patients in use of anticoagulants
* Known thrombophilia
* Presence of saphenous vein tortuosity and/or depth less then 7 mm from the skin
* GSV diameter < 5mm and > 12 mm
* Previous deep vein thrombosis
* Peripheral arterial disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-06 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
GSV occlusion | 3 months
  GSV occlusion verified by blinded DS operator
GSV occlusion | 6 months
  GSV occlusion verified by blinded DS operator

SECONDARY OUTCOMES:
Pain VAS | 1 week
  Pain VAS by blinded Outcomes Assessor
Post operative bruising | 1 week
  The bruised area traced manually, and the surface area estimated by placing the tracing on a square chart.
  Assessment by blinded Outcomes Assessor.
Post operative sensory abnormality | 1 week
  Overall incidence of postoperative sensory abnormality: Numbness or decreased sensation, paresthesia and dysesthesia.
  Assessment by blinded Outcomes Assessor
Venous Clinical Severity Score (VCSS) | 6 months
  Difference from baseline. Assessment by blinded Outcomes Assessor.
Aberdeen Varicose Vein Questionnaire (AVVQ) | 6 months
  Difference from baseline. Assessment by blinded Outcomes Assessor.
Deep Venous Thrombosis (DVT) | 1 week
  Presence of DVT verified by blinded DS operator
Clinical Etiology Anatomy Pathophysiology (CEAP) | 6 months
  Difference from baseline. Assessment by blinded Outcomes Assessor.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio H Rossi, PHD, Principal Investigator — Dante Pazzanese
Locations (1):
- Instituto Dante Pazzanese de Cardilogia, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rossi FH, Beteli CB, Zamorano MB, Silva LM. Immediate effects of endovascular electrocauterization in lower limb varicose veins. J Vasc Bras 11(3): 305-309, 2012.
- [Background] Rossi FH, Izukawa NM, Silva DG, Chen J, Prakasan AK, Zamorano MM, Silva LM. Effects of electrocautery to provoke endovascular thermal injury. Acta Cir Bras. 2011 Oct;26(5):329-32. doi: 10.1590/s0102-86502011000500001. PMID 21952653
- See also: free article — http://www.scielo.br/pdf/acb/v26n5/a01v26n5.pdf
- See also: free article — http://www.scielo.br/pdf/jvb/v11n4/09.pdf